CLINICAL TRIAL: NCT01084408
Title: Randomized Trial on the Treatment of Coronary De-novo Lesions With a Drug Eluting Stent or a Drug Coated Balloon
Brief Title: Efficacy of the SeQuent®Please in the Treatment of De-novo Stenoses Versus Taxus™Liberté™
Acronym: PEPCAD-DEBonly
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: no suitable patients
Sponsor: University Hospital, Saarland (Other)
Responsible Party: Principal Investigator, Bruno Scheller, MD, University Hospital, Saarland
Organization: Universität des Saarlandes (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pac 14
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Coronary De-novo Stenoses
Keywords: de-novo; coronary stenoses; PEPCAD; DEBonly; Paclitaxel
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequent®Please (Active Comparator)
  Interventions: Device: SeQuent®Please (Paclitaxel coated balloon)
- Taxus™Liberté™ (Active Comparator)
  Interventions: Device: Taxus™Liberté™ (Paclitaxel eluting stent)

INTERVENTIONS:
Device: SeQuent®Please (Paclitaxel coated balloon) — PCI of de-novo lesions
  Arms: Sequent®Please
Device: Taxus™Liberté™ (Paclitaxel eluting stent) — PCI of de-novo lesions
  Arms: Taxus™Liberté™

SUMMARY:
The aim of the trial is to assess the efficacy of the Paclitaxel-coated SeQuent®Please angioplasty balloon in the treatment of stenoses in native coronary arteries compared to a drug eluting stent.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Clinical evidence of stable or unstable angina or a positive functional study
* Single, stenotic de novo lesion in a native coronary artery, type A or selected B1 (see 4.3.1.1 Definition of lesion types)
* Diameter stenosis > 70% (visual estimate)
* Vessel diameter 2.5 - 3.5 mm
* Female patients can enter this study if they are post-menopausal for at least two years or have undergone hysterectomy or sterilization
* Signed patient informed consent form
* Patient's and treating physician's agree that the patient will return for all required post procedure follow-up assessments as defined in the clinical protocol

Exclusion Criteria:

* Left ventricular ejection fraction of < 30%
* Visible thrombus proximal to the lesion
* Expection that treatment with devices other than PTCA will be required for this lesion.
* Stenosis is within a bypass graft
* Known hypersensitivity or contraindication to aspirin, heparin, clopidogrel, paclitaxel, or a sensitivity to contrast media which cannot be adequately pre-medicated
* Other medical illness (i.e. cancer, liver disease or congestive heart failure) that may require cytostatic or radiation therapy, cause the subject to be non-compliant with the protocol, confound the data interpretation or is associated with limited life-expectancy (i.e., less than two years).
* Acute myocardial infarction within the past 72 hours of the intended treatment (de-fined as: Q wave infarction having total creatinine kinase (CK) >3 times the upper normal limit, or CK remains elevated above hospital normal at time of treatment)
* Chronic renal insufficiency with serum creatinine > 2.0 mg%
* Significant gastrointestinal (GI) bleed within the past six months.
* History of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Extensive peripheral vascular disease that precludes safe 6 French sheath insertion and / or requires additional anti-platelet and / or anti-coagulation treatment.
* Participating in another device or drug study within the last 6 months which may inter-fere with the interpretation of results of this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-03-01 (Actual); Primary Completion 2012-03-01 (Actual); Study Completion 2013-03-01 (Actual)

PRIMARY OUTCOMES:
Late lumen loss | 6 months
  Late lumen loss = MLD in-lesion initially - MLD in lesion after six months (after nitroglycerin in identical projections); assessment by an independent Core Lab.

SECONDARY OUTCOMES:
Thrombotic occlusion of the target lesion | 30 days, 6, 12, 24, 60 months
Revascularization of the target lesion | 30 days, 6, 12, 24, 60 months
Myocardial infarction | 30 days, 6, 12, 24, 60 months
Death | 30 days, 6, 12, 24, 60 months
Combined clinical endpoint (MACE) | 30 days, 6, 12, 24, 60 months
  consisting of thrombotic occlusion of the treated segment, target lesion revascularization, myocardial infarction, or death

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Scheller, Prof. Dr. med, Principal Investigator — Uniklinikum des Saarlandes
Locations (2):
- Germany (2):
  - Klinik für Kardiologie, Angiologie und Konservative Intensivtherapie Klinikum Ernst von Bergmann, Postdam, Brandenburg
  - Medizinisches Versorgungszentrum, Hamburg